CLINICAL TRIAL: NCT02426515
Title: Cryotherapy to Improve Outcomes in Lower Third Molar Surgery
Acronym: COOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Birmingham Community Healthcare NHS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-080
Record Dates: First submitted 2015-04-17; First posted 2015-04-27 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Oral Surgery
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hilotherm® Device (Experimental): Patients undergo removal of lower third molar with Hilotherm® cooling device applied.
  Interventions: Device: Hilotherm® cooling device and face mask
- Control (No Intervention): Patients undergo removal of lower third molar without the Hilotherm® cooling device applied.

INTERVENTIONS:
Device: Hilotherm® cooling device and face mask — Hilotherm® is an external cooling device and facial mask through which water circulates at a controlled temperature This allows continuous cooling of the face, and is thought to reduce post-operative swelling and pain.
  Arms: Hilotherm® Device

SUMMARY:
This study is looking to see whether cooling the face using a special cooling device (Hilotherm®) before and during the removal of wisdom teeth will reduce the pain and discomfort patients feel after the procedure. The surgical removal of lower third molars (wisdom teeth) is arguably the most commonly performed surgical procedure worldwide. If this study shows that application of cold before and throughout the procedure is a simple way to reduce post-operative symptoms, it could benefit thousands of patients every year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18+ years requiring surgical removal of a single (unilateral) mandibular wisdom tooth
2. Tooth requiring full mucoperiosteal flap and bone removal for removal of tooth
3. Written informed consent

Exclusion Criteria:

1. Patients refusing to give written informed consent
2. Clinically significant or unstable physical or mental disability rendering the participants incapable of complying with the study protocol as judged by the investigator
3. Pregnant women
4. Patients taking long-term anti-microbial or anti-inflammatory drugs
5. Patients requiring pre-operative antibiotics for surgery
6. Patients requiring concomitant extractions or contralateral lower 3rd molar removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 7 days
  Post operative pain 7 days after operation as measured in mm from VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham Dental Hospital, Birmingham, United Kingdom